CLINICAL TRIAL: NCT01743625
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-Controlled, Parallel-Group Evaluation of the Safety and Analgesic Efficacy of COV155 Tablets in Moderate to Severe Post-Operative Bunionectomy Pain Followed by an Open-Label Extension
Brief Title: Safety and Efficacy Study of COV155 for Post-operative Bunionectomy Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COV15010232
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Pain, Postoperative; Bunion
MeSH Terms: conditions — Pain, Postoperative; Bunion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- COV155 (Experimental): COV155, loading dose of 3 tablets followed by 2 tablets every 12 hours for 48 hours.
  Interventions: Drug: COV155
- Placebo (Placebo Comparator): Matching tablet to COV155 without containing active ingredients, loading dose of 3 tablets followed by 2 tablets every 12 hours for 48 hours.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: COV155 — COV155 tablets
  Other Names: MNK155
  Arms: COV155
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to show the effectiveness of COV155 compared to placebo in subjects with acute moderate to severe pain following bunionectomy surgery.

ELIGIBILITY:
Inclusion Criteria

* Voluntarily provide written informed consent
* General good health
* 18 to 75 years of age
* Scheduled for primary unilateral first metatarsal bunionectomy (with no collateral procedures)
* Body mass index ≤33
* Female subjects eligible if

  * Not pregnant or lactating; not planning to become pregnant for duration of study;
  * Surgically sterile, or have a monogamous partner who is surgically sterile, or at least 2 years postmenopausal, or practicing acceptable birth control for more than 2 months prior to Screening, during the study and for 1 week following last dose of COV155
* Male subjects must be sterile (biologically or surgically) or use reliable birth control during the study until at least 1 week after the last dose of COV155
* Classified as either Physical Status-1 (PS) or PS-2 by the American Society of Anesthetists (ASA) Physical Status Classification System.
* Willing to complete pain assessments and clinic visits.
* Additional inclusion criterion for randomization into the Double-Blind Phase: Subjects must experience postoperative pain intensity score ≥5 on a 0 to 10 Numerical Pain Rating Score (NPRS) more than 1 hour, and less than 9 hours after discontinuing the nerve block, and at least 30 minutes after the last ice pack has been removed (if used).

Exclusion Criteria

* Uncontrolled medical condition, serious intercurrent illness, clinically significant general health condition, or extenuating circumstance that may significantly decrease study compliance or otherwise preclude study participation
* Clinically significant abnormal ECG at Screening
* Gastric bypass surgery or gastric band
* Previous abdominal surgery within the past year or history of abdominal adhesions, known or suspected paralytic ileus
* History of any medical condition that would alter the absorption, distribution, metabolism or excretion of COV155 including but not limited to severe chronic diarrhea, chronic constipation, severe irritable bowel syndrome, or unexplained weight loss
* History of severe bronchial asthma, hypercarbia, hypoxia or sleep apnea
* Certain lab abnormalities
* Addison's disease, benign prostatic hyperplasia, or kidney disease
* Donated blood or blood components within 3 months prior to Screening or during study
* Known allergy/hypersensitivity to any opioid analgesics, anesthetics, acetaminophen, non steroidal anti-inflammatory drugs (NSAIDs)
* History of intolerance to short term opioid use
* Unable to discontinue the use of prohibited medications or a history of substance or alcohol abuse within 2 years prior to Screening or a positive quantitative urine drug test at Screening
* Positive for human immunodeficiency virus, hepatitis B or C
* Dysphagia and/or cannot swallow study treatment whole
* History of migraine or frequent headaches within the previous 2 years, seizures, or are currently taking anticonvulsants
* Previously received COV155 in a clinical study, or undergone a bunionectomy within the last 3 months
* Received any investigational drugs or devices within 4 weeks prior to Screening or during study
* Active malignancy or history of malignancy within 2 years prior to Screening, other than completely eradicated cervical squamous cell carcinoma in situ or basal skin cancer
* Currently taking neuroleptics or stable doses of a benzodiazepine
* Other criteria as specified in the protocol
* Additional exclusion criterion for randomization into the Double-Blind Phase: Have surgical complications that could compromise the safety of the subject or confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
SPID48 (Summed pain intensity difference) | 48 hours
  48 hour Summed pain intensity difference

SECONDARY OUTCOMES:
Safety and tolerability of COV155 | 48 hours
  Safety and tolerability to be evaluated with physical exams, vital signs, pulse oximetry, clinical laboratory tests, electrocardiograms, and adverse events
Onset of analgesia of COV155 versus placebo | 48 hours
  Onset of confirmed perceptible pain relief, time to meaningful pain relief, and time to peak pain intensity difference
Analgesic effects of COV155 versus placebo | 48 hours
  Pain intensity scores, pain intensity differences, and summed pain intensity differences; pain relief scores and total pain relief; percent responders; mean dosing interval; use of rescue medication; global assessment of subject satisfaction with study treatment.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Anaheim Clinical Trials, Anaheim, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - Chesapeake Research Group, LLC, Pasadena, Maryland
  - Endeavor Clinical Trails, PA, San Antonio, Texas
  - Jean Brown Research, Inc., Salt Lake City, Utah